CLINICAL TRIAL: NCT06408935
Title: A Phase 3b, Open-label, Multicenter Study to Evaluate Transmural Healing and Disease Modifying Effect of Guselkumab in Crohn's Disease Patients
Brief Title: Transmural Healing and Disease-Modifying Effect of Guselkumab in Crohn's Disease Patients
Acronym: REASON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNTO1959CRD3008; CNTO1959CRD3008 (Other: Janssen Research & Development, LLC); 2023-504040-34-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Guselkumab (Experimental): Participants will receive guselkumab 200 milligram (mg) intravenously (IV) at week 0, 4 and 8. Afterwards, participants will be alternately assigned at study level to 2 dose cohorts, high dose (200 mg subcutaneous (SC) every 4 weeks (Q4W) starting at week 12) through week 92 or low dose (100 mg SC every 8 weeks (Q8W) starting at week 16) through week 88. Starting at Week 24, participants in the low-dose cohort will be permitted to escalate to the 200 mg SC Q4W regimen if they are symptomatic and at the discretion of the investigator.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered IV and SC.
  Other Names: CNTO1959; TREMFYA

SUMMARY:
The purpose of this study is to evaluate the efficacy of guselkumab in healing of all layers of the digestive tract (transmural healing) with the help of a score called Magnetic Resonance Index of Activity (MaRIA) based on a scan at Week 48.

ELIGIBILITY:
Inclusion Criteria:

* Has luminal Crohn's disease (CD) of at least 3 months duration (defined as a minimum of 12 weeks), with colitis, ileitis, or ileocolitis, confirmed at any time in the past by radiography, histology, and/or endoscopy
* Has clinically active CD, defined as a baseline CD activity index (CDAI) score greater than or equal to (>=)220 but <=450 and either: a. Mean daily stool frequency (SF) count >=4, based on the unweighted CDAI component of the number of liquid or very soft stools or b. Mean daily AP score >=2, based on the unweighted CDAI component of abdominal pain (AP)
* Active transmural activity in at least one segment (segmental magnetic resonance index of activity [MaRIA] >= 11)
* a. Has demonstrated inadequate response/intolerance to conventional therapy; b. Has previously demonstrated lack of initial response (that is, primary non-responders), responded initially but then lost response with continued therapy (that is, secondary non-responders), or was intolerant to a maximum of 1 class of advanced therapies at a dose approved for the treatment of Crohn's disease (that is, janus kinase [JAK] inhibitors, infliximab, adalimumab, certolizumab pegol, vedolizumab, ustekinumab, or approved biosimilars for these agents)

Exclusion Criteria:

* Has complications of Crohn's disease, such as symptomatic strictures or stenoses (unless less than [<]3 centimeter (cm) dilatation and not symptomatic or displaying associated fistula/fistulae and/or or abscess), fibrotic stenosis, internal fistulas, short gut syndrome, or any other manifestation, that might be anticipated to require surgery, could preclude the use of the CDAI to assess response to therapy, or would possibly confound the ability to assess the effect of treatment with guselkumab
* Currently has or is suspected to have an abscess. Recent cutaneous and perianal abscesses are not exclusionary if drained and adequately treated at least 3 weeks before baseline, or 8 weeks before baseline for intra-abdominal abscesses, provided that there is no anticipated need for any further surgery. Participants with active perianal fistulas may be included if there are no associated stenoses, no anticipated surgery and no abscesses currently identified
* Has had any kind of bowel resection within 6 months, or any other intra-abdominal or other major surgery within 12 weeks before baseline
* Has a draining (that is, functioning) stoma or ostomy
* Has a stool culture or other examination positive for an enteric pathogen, including Clostridioides difficile (formerly known as Clostridium difficile) toxin, in the previous 4 months, unless a repeat examination is negative and there are no signs of ongoing infection with that pathogen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-06-08 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Magnetic Resonance Index of Activity (MaRIA) Less Than (<)11 in All Intestinal Segments at Week 48 | At Week 48
  Percentage of participants achieving a MaRIA <11 in all intestinal segments at Week 48 will be reported. The MaRIA scoring system is used to grade severity in Crohn's Disease (CD) by assessing ileocolonic CD activity on contrast-enhanced magnetic resonance imaging (MRI) enterography. Active disease is defined as a MaRIA score greater than or equal to (>=)7 whereas severe disease is defined as a MaRIA score >=11.

SECONDARY OUTCOMES:
Percentage of Participants Achieving a MaRIA <11 in All Intestinal Segments at Weeks 16 and 96. | At Weeks 16 and 96
  Percentage of participants achieving a MaRIA <11 in all intestinal segments at Weeks 16 and 96 will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic CD activity on contrast-enhanced MRI enterography. Active disease is defined as a MaRIA score >=7 whereas severe disease is defined as a MaRIA score >=11.
Percentage of Participants Achieving a MaRIA <11 and a Reduction of >=5 Points From Baseline in All Segments at Weeks 16, 48, and 96 | At Weeks 16, 48, and 96
  Percentage of participants achieving a MaRIA <11 and a reduction of >=5 points from baseline in all segments at Weeks 16, 48, and 96 will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic Crohn disease activity on contrast-enhanced MRI enterography. Active disease is defined as a MaRIA score >=7 whereas severe disease is defined as a MaRIA score >=11.
Percentage of Participants Achieving a MaRIA <11 in All Segments and Endoscopic Remission at Weeks 48 and 96 | At Week 48 and 96
  Percentage of participants achieving a MaRIA <11 in all segments and endoscopic remission at Weeks 48 and 96 will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic CD activity on contrast-enhanced MRI enterography. Active disease is defined as a MaRIA score >=7 whereas severe disease is defined as a MaRIA score >=11. Endoscopic remission is defined as simple endoscopic score for Crohn's Disease (SES-CD) total score <=4 with at least 2 points reduction from baseline and no sub-score >1 in any individual component.
Percentage of Participants Achieving a MaRIA <11 in All Segments and Endoscopic Response at Weeks 48 and 96. | At Weeks 48 and 96
  Percentage of participants achieving a MaRIA <11 in all segments and endoscopic response at Weeks 48 and 96 will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic CD activity on contrast-enhanced MRI enterography. Active disease is defined as a MaRIA score >=7 whereas severe disease is defined as a MaRIA score >=11. Endoscopic Response is defined as >=50% improvement from baseline in simple endoscopic score for Crohn's Disease (SES-CD) total score or SES-CD total score <=2.
Percentage of Participants Achieving a MaRIA <11 in All Segments, Patient-Reported Outcome-2 (PRO-2) Remission, and No Worsening of Abdominal Pain (AP) or Stool Frequency (SF) From Baseline | At Weeks 16, 48 and 96
  Percentage of participants achieving a MaRIA <11 in all segments and PRO-2 remission and no worsening of abdominal pain (AP) or stool frequency (SF) from baseline will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic CD activity on contrast-enhanced MRI enterography. Active disease is defined as a MaRIA score greater than or equal to (>=)7 whereas severe disease is defined as a MaRIA score >=11. PRO-2 remission is defined as defined as AP mean daily score <=1 and a SF mean daily score <=3, and no worsening of AP or SF from baseline.
Percentage of Participants Achieving a MaRIA <11 in All Segments and Biomarkers Remission | At Weeks 16, 48 and 96
  Percentage of participants achieving a MaRIA <11 in all segments and biomarkers remission will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic CD activity on contrast-enhanced MRI enterography. Active disease is defined as a MaRIA score >=7 whereas severe disease is defined as a MaRIA score >=11. Biomarker remission is defined as CRP <=3 mg/L and fecal calprotectin (fCal) <=250 mcg/g.
Percentage of Participants Achieving a MaRIA <11 in All Segments, PRO-2, and Endoscopic Remission | At Weeks 48 and 96
  Percentage of participants achieving a MaRIA <11 in all segments, PRO-2, and endoscopic remission will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic CD activity on contrast-enhanced MRI enterography. The MaRIA scale is based on features that are predictors for active disease; bowel wall thickness, presence of mucosal ulcers, presence of mural edema, measurement of WSI before and after IV contrast administration and RCE of the intestinal wall. Active disease is defined as a MaRIA score greater than or equal to (>=)7 whereas severe disease is defined as a MaRIA score >=11. PRO is defined as defined as AP mean daily score <=1 and a SF ) mean daily score <=3, and no worsening of AP or SF from baseline. Endoscopic remission is defined as SES-CD total score <=4 with at least 2 points reduction from baseline and no sub-score >1 in any individual component.
Percentage of Participants Achieving a MaRIA <7 in All Intestinal Segments at Weeks 16, 48 and 96 | At Weeks 16, 48 and 96
  Percentage of participants achieving a MaRIA <7 in all intestinal segments at Weeks 16, 48 and 96 will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic Crohn disease activity on contrast-enhanced MRI enterography. Active disease is defined as a MaRIA score >=7 whereas severe disease is defined as a MaRIA score >=11.
Percentage of Participants Achieving a MaRIA <7 in All Segments and Endoscopic Remission at Weeks 48 and 96 | At Weeks 48 and 96
  Percentage of participants achieving a MaRIA <7 in all segments and endoscopic remission at Weeks 48 and 96 will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic CD activity on contrast-enhanced MRI enterography. Active disease is defined as a MaRIA score greater than or equal to (>=)7 whereas severe disease is defined as a MaRIA score >=11. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic Crohn disease activity on contrast-enhanced MRI enterography. The MaRIA scale is based on features that are predictors for active disease; bowel wall thickness, presence of mucosal ulcers, presence of mural edema, measurement of WSI before and after IV contrast administration and RCE of the intestinal wall. Active disease is defined as a MaRIA score greater than or equal to (>=)7 whereas severe disease is defined as a MaRIA score >=11.
Absolute Value of Global Simple MaRIA Score Through Week 96 | Baseline up to Week 96
  Absolute Value of global simple MaRIA score through Week 96 will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic Crohn disease activity on contrast-enhanced MRI enterography. Active disease is defined as a MaRIA score greater than or equal to (>=)7 whereas severe disease is defined as a MaRIA score >=11.
Change From Baseline in the Global Simple MaRIA Score Through Week 96 | Up to Week 96
  Change from baseline in the global simple MaRIA score through Week 96 will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic CD activity on contrast-enhanced MRI enterography. Active disease is defined as a MaRIA score >=7 whereas severe disease is defined as a MaRIA score >=11.
Percentage of Participants Achieving a MaRIA <7 in All Intestinal Segments and Not Receiving Corticosteroids at Weeks 16, 48, and 96 | At Weeks 16, 48, and 96
  Percentage of participants achieving a MaRIA <7 in all intestinal segments and not receiving corticosteroids at Weeks 16, 48, and 96 will be reported. The MaRIA scoring system is used to grade severity in CD by assessing ileocolonic CD activity on contrast-enhanced MRI enterography. Active disease is defined as a MaRIA score >=7 whereas severe disease is defined as a MaRIA score >=11.
Percentage of Participants Achieving Transmural Segmental Response with Intestinal Ultrasound (IUS) at Weeks 4, 8, 16, 48, and 96 | Baseline, at Weeks 4, 8, 16, 48, and 96
  Percentage of participants achieving transmural segmental response with IUS at Weeks 4, 8, 16, 48, and 96 will be reported. Transmural segmental response with IUS is defined as a reduction from baseline of 25 percent (%) in BWT or a reduction from baseline of bowel wall thickness (BWT) >=2 mm or a reduction from baseline of BWT >=1 millimeter (mm) plus a decrease from baseline in color doppler signal (CDS) >=1 point.
Percentage of Participants with Transmural Response (total) at Weeks 4, 8, 16, 48, and Week 96 | Baseline, at Weeks 4, 8, 16, 48, and Week 96
  Percentage of participants with transmural response (total) at Weeks 4, 8, 16, 48, and Week 96 will be reported. Transmural segmental response with IUS is defined as: a reduction from baseline of 25 percent (%) in BWT or a reduction from baseline of BWT >=2 millimeter (mm) or a reduction from baseline of BWT >=1 mm plus a decrease from baseline in color doppler >=1 point, per baseline pathological segment. Transmural response (total) requires that at least one pathological segment at baseline fulfills the criteria.
Percentage of Participants Achieving Transmural Remission with IUS at Weeks 4, 8, 16, 48, and 96 | At Weeks 4, 8, 16, 48, and 96
  Percentage of participants achieving transmural remission with IUS at Weeks 4, 8, 16, 48, and 96 will be reported. Transmural remission with IUS is defined as BWT <=3 mm for ileum and colon plus color doppler signal 0, in all segments.
Absolute Value of International Bowel Ultrasound Segmental Activity Score (IBUS-SAS) Through Week 96 | Baseline up to Week 96
  Absolute value of IBUS-SAS through Week 96 will be reported. IBUS-SAS score is defined as 4*BWT+15*IMF+7*CDS+4*BWS.
Change from Baseline in International Bowel Ultrasound Segmental Activity Score (IBUS-SAS) Through Week 96 | Up to Week 96
  Change from baseline in IBUS-SAS through Week 96 will be reported. IBUS-SAS score is defined as 4*BWT+15*IMF+7*CDS+4*BWS.
Percentage of Participants Achieving IBUS-SAS Response at Weeks 4, 8, 16, 48, and Week 96 | Baseline, at Weeks 4, 8, 16, 48, and Week 96
  Percentage of participants achieving IBUS-SAS response at Weeks 4, 8, 16, 48, and Week 96 will be reported. IBUS-SAS is defined as a reduction in IBUS-SAS score from baseline of >=10 points per baseline pathological segment and segmental score <=12 (if not pathological), at baseline.
Percentage of Participants Achieving BWT <=3 mm for Ileum and Colon Plus CDS 0, in all segments and Participants Not Receiving Corticosteroids at Weeks 4, 8, 16, 48, and 96 | At Weeks 4, 8, 16, 48, and 96
  Percentage of participants achieving BWT <=3 mm for Ileum and Colon plus CDS 0, in all segments at Weeks 4, 8, 16, 48, and 96 will be reported. Participants not receiving corticosteroids achieving BWT <=3 mm for Ileum and Colon plus CDS 0 at Weeks 4, 8, 16, 48, and 96 will be reported.
Absolute Value of BWT through Week 96 | Baseline up to Week 96
  Absolute Value of BWT through Week 96 will be reported.
Change From Baseline in BWT Through Week 96 | Up to Week 96
  Change from baseline in BWT through Week 96 will be reported.
Absolute Value of Simple IUS Score For CD (SUS-CD) Score Through Week 96 | Baseline up to Week 96
  Absolute value of SUS-CD score through Week 96 will be reported. SUS-CD is based on the sum of classifications for BWT and CDS for all segments.
Change From Baseline in the SUS-CD Score Through Week 96 | Up to Week 96
  Change from Baseline in the SUS-CD score through Week 96 will be reported. SUS-CD is based on the sum of classifications for BWT and CDS for all segments.
Percentage of Participants Achieving Endoscopic Response at Weeks 48 and 96 | Weeks 48 and 96
  Percentage of participants with transmural response (total) at Weeks 48 and Week 96 will be reported. Endoscopic Response is defined as >=50% improvement from baseline in SES-CD total score or SES-CD <=2.
Percentage of Participants Achieving Endoscopic Remission at Weeks 48 and 96 | At Weeks 48 and 96
  Percentage of participants achieving endoscopic remission at Weeks 48 and 96 will be reported. Endoscopic remission is defined as SES-CD total score <=4 with at least 2 points reduction from baseline and no sub-score >1 in any individual component.
Absolute Value of SES-CD Total Score Through Week 96 | Baseline up to Week 96
  Absolute value of SES-CD total score through Week 96 will be reported. The SES-CD score is used to evaluate endoscopic improvement. The SES-CD is based on the evaluation of 4 endoscopic components (presence/size of ulcers, proportion of mucosal surface covered by ulcers, proportion of mucosal surface affected by any other lesions, and presence/type of narrowing/strictures) across 5 ileocolonic segments. An overall total SES-CD score is derived from the sum of all the component scores and can range from 0 to 56.
Change From Baseline in the SES-CD Total Score Through Week 96 | Up to Week 96
  Change from baseline in the SES-CD total score through Week 96 will be reported. The SES-CD score is used to evaluate Endoscopic Improvement. The SES-CD is based on the evaluation of 4 endoscopic components (presence/size of ulcers, proportion of mucosal surface covered by ulcers, proportion of mucosal surface affected by any other lesions, and presence/type of narrowing/strictures) across 5 ileocolonic segments. An overall total SES-CD score is derived from the sum of all the component scores and can range from 0 to 56.
Percentage of Participants (Not Receiving Corticosteroids) Achieving Endoscopic Remission at Weeks 48 and 96 | Baseline, at Weeks 48 and 96
  Percentage of participants (not receiving corticosteroids) achieving endoscopic remission at Weeks 48 and 96 will be reported. Endoscopic remission is defined as SES-CD total score <=4 with at least 2 points reduction from baseline and no sub-score >1 in any individual component.
Percentage of Participants Achieving Endoscopic Healing of the Intestinal Mucosa at Weeks 48 and 96 | At Weeks 48 and 96
  Percentage of participants achieving endoscopic healing of the intestinal mucosa at Weeks 48 and 96 will be reported. Endoscopic healing is defined as the resolution (absence) of mucosal ulcers in response to a therapeutic intervention.
Percentage of Participants Achieving Crohn's Disease Activity Index (CDAI) <150 at Weeks 4, 8, 16, 48 and 96 | At Weeks 4, 8, 16, 48 and 96
  Percentage of participants achieving CDAI <150 at Weeks 4, 8, 16, 48 and 96 will be reported. CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid or very soft stools, abdominal pain (AP)/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. The last 4 variables are scored over 7 days by the participant on a diary card that participants are to complete on daily basis.
Percentage of Participants Achieving a Reduction in the CDAI Score of >=100 points or CDAI <150 From Baseline at Weeks 4, 8, 16, 48, and 96 | At Weeks 4, 8, 16, 48, and 96
  Percentage of participants achieving a reduction in the CDAI score of >=100 points or CDAI <150 from Baseline at Weeks 4, 8, 16, 48, and 96 will be reported. CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid or very soft stools, abdominal pain (AP)/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. The last 4 variables are scored over 7 days by the participant on a diary card that participants are to complete on daily basis.
Percentage of Participants (Not Receiving Corticosteroids) Achieving CDAI Score <150 at Weeks 4, 8, 16, 48 and 96 | At Weeks 4, 8, 16, 48 and 96
  Percentage of participants (not receiving corticosteroids) achieving CDAI Score <150 at Weeks 4, 8, 16, 48 and 96 will be reported. CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid or very soft stools, abdominal pain (AP)/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. The last 4 variables are scored over 7 days by the participant on a diary card that participants are to complete on daily basis.
Absolute Value of CDAI Score Through Week 96 | Baseline up to Week 96
  Absolute Value of CDAI score through Week 96 will be reported. CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid or very soft stools, abdominal pain (AP)/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. The last 4 variables are scored over 7 days by the participant on a diary card that participants are to complete on daily basis.
Change From Baseline in CDAI Score Through Week 96 | Up to Week 96
  Change from baseline in CDAI score through Week 96 will be reported. CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid or very soft stools, abdominal pain (AP)/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. The last 4 variables are scored over 7 days by the participant on a diary card that participants are to complete on daily basis.
Percentage of Participants Achieving PRO-2 Remission at Weeks 4, 8, 16, 48, and Week 96 | At Weeks 4, 8, 16, 48, and Week 96
  Percentage of participants achieving PRO-2 remission at Weeks 4, 8, 16, 48, and Week 96 will be reported. PRO-2 remission is defined as AP mean daily score <=1 and a SF mean daily score <=3, and no worsening of AP or SF from baseline.
Percentage of Participants Achieving Inflammatory Bowel Disease Questionnaire (IBDQ) Remission at Weeks 48 and 96 | At Week 48 and Week 96
  Percentage of participants achieving IBDQ remission at Weeks 48 and 96 will be reported. The IBDQ is a validated, 32-item, self-reported questionnaire for participants with IBD to evaluate PROs across 4 dimensions: bowel symptoms (loose stools, AP), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability).
Percentage of Participants Achieving IBDQ Response at Weeks 48 and 96 | Baseline, at Weeks 48 and 96
  Percentage of participants achieving IBDQ response at Weeks 48 and 96 will be reported. IBDQ response is defined as >=16-point improvement in IBDQ score from baseline. IBDQ score ranges from 32 to 224, with higher scores indicating better outcomes.
Absolute Value of IBDQ Through Week 96 | Baseline up to Week 96
  Absolute value of IBDQ through Week 96 will be reported. The IBDQ is a validated, 32-item, self-reported questionnaire for participants with IBD to evaluate PROs across 4 dimensions: bowel symptoms (loose stools, AP), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Scores range from 32 to 224, with higher scores indicating better outcomes.
Change From Baseline in IBDQ Score Through Week 96 | Up to Week 96
  Change from baseline in IBDQ score through Week 96 will be reported. The IBDQ is a validated, 32-item, self-reported questionnaire for participants with IBD to evaluate PROs across 4 dimensions: bowel symptoms (loose stools, AP), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Scores range from 32 to 224, with higher scores indicating better outcomes.
Change from Baseline in Urgency Numeric Rating Scale (UNRS) Through Week 96 | Baseline up to Week 96
  Change from baseline in UNRS through Week 96 will be reported. UNRS is designed to assess changes in the severity of bowel urgency (sudden or immediate need). Severity of bowel urgency is defined by the patient's perception of overall experience in which respondents consider the immediacy of bowel movement urgency severity over 24 h on an 11-point horizontal NRS ranging from 0 ('no urgency') to 10 ('worst possible urgency').
Percentage of Participants Achieving C-reactive Protein (CRP) Normalization at Weeks 4, 8, 16, 48, and Week 96 | Baseline, at Weeks 4, 8, 16, 48, and Week 96
  CRP normalization is defined as CRP <=3 mg/L, among participants with baseline elevation in CRP (that is, >3 mg/L).
Percentage of Participants Achieving >=50% Improvement of CRP Response From Baseline at Weeks 4, 8, 16, 48, and 96 | Baseline, at Weeks 4, 8, 16, 48, and 96
  Percentage of participants achieving >=50% improvement of CRP response from baseline at Weeks 4, 8, 16, 48, and 96 will be reported.
Percentage of Participants Achieving fCal Normalization at Weeks 4, 8, 16, 48, and 96 | Baseline, at Weeks 4, 8, 16, 48, and 96
  Percentage of participants achieving fCal normalization at Weeks 4, 8, 16, 48, and 96 will be reported. fCal normalization is defined as fCal <=250 mcg/g among participants with elevated fCal at baseline.
Percentage of Participants Achieving >=50% Improvement of fCal Response From Baseline at Weeks 4, 8, 16, 48, and 96 | Baseline, at Weeks 4, 8, 16, 48, and 96
  Percentage of participants achieving >=50% improvement of fCal response from baseline at Weeks 4, 8, 16, 48, and 96 will be reported.
Change From Baseline in CRP and fCal Levels Over Time | Baseline, Weeks 4, 8, 16, 32, 48, and 96
  Change from baseline in CRP and fCal levels over time will be reported.
Values of CRP and fCal Levels Over Time | Baseline, Weeks 4, 8, 16, 32, 48, and 96
  Values of CRP and fCal levels over time will be reported.
Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TSAEs) Through Week 48 | Up to Week 48
  An AE is any untoward medical occurrence in a clinical study subject administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as the AEs occurring after first administration of study intervention (or worsened since then). An serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product. TESAEs are defined as serious events between administration of study drug and after the last dose that were absent before treatment or that worsen relative to pretreatment state.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Cilag Ltd. Clinical trial, Study Director — Janssen-Cilag Ltd.
Locations (83):
- United States (4):
  - Center for Colitis and Crohns Disease University of California, San Francisco, California
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - Washington University School Of Medicine, St Louis, Missouri
  - Medical University of South Carolina, Charleston, South Carolina
- Australia (5):
  - The Queen Elizabeth Hospital, Adelaide
  - Concord Repatriation General Hospital, Concord
  - Northern Hospital, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Mater Hospital Brisbane, South Brisbane
- Belgium (3):
  - AZ Maria Middelares, Ghent
  - CHU de Liege, Liège
  - Vitaz, Sint-Niklaas
- Brazil (4):
  - Cliged, Macaé
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - NPCRS Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre
  - INTEGRAL Pesquisa e Ensino, Votuporanga
- Canada (3):
  - Foothills Hospital, Calgary, Alberta
  - Western University & London Health Sciences Centre, London, Ontario
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
- Czechia (3):
  - Nemocnice Ceske Budejovice a s, České Budějovice
  - Hepato-gastroenterologie HK, s.r.o., Hradec Králové
  - ISCARE a.s., Prague
- France (6):
  - CHU Amiens Picardie, Amiens
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Aphm - Hopital Nord, Marseille
  - CHU de Nantes hotel Dieu, Nantes
  - APHP - Hopital Bichat - Claude Bernard, Paris
- Germany (13):
  - Klinikum Augsburg, Augsburg
  - Charite Universitaetsmedizin Berlin, Berlin
  - Praxis Fur Gastroenteroligie, Berlin
  - Medizinisches Versorgungszentrum (MVZ) Dachau, Dachau
  - Universitatsklinikum Frankfurt/ Medizinische Klinik 1, Frankfurt
  - Universitatsmedizin Gottingen, Göttingen
  - BSF Studiengesellschaft, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Schleswig Holstein, Kiel
  - Staedtisches Klinikum Lueneburg, Lüneburg
  - MVZ Portal 10, Münster
  - Siloah St Trudpert Klinikum, Pforzheim
  - Universitaetsklinikum Ulm, Ulm
- Israel (7):
  - Rambam Medical Center, Haifa
  - The Edith Wolfson Medical Center, Holon
  - Hadassah Medical Organization, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (11):
  - Azienda Ospedaliera Policlinico S. Orsola-Malpighi, Bologna
  - ASST Fatebenefratelli Sacco, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Universita Di Napoli Federico Ii, Napoli
  - ASL Toscana Nord Ovest PO Valdera Ospedale Lotti, Pontedera Pisa
  - Asst Rhodense - Ospedale Di Rho, Rho
  - Universita Campus Bio-Medico di Roma, Roma
  - Fondazione Policlinico Tor Vergata, Roma
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - IRCCS Humanitas Rozzano-IBD Center Malattie Infiammatorie Croniche Intestinali, Rozzano
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Poland (8):
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Centrum Medyczne Medyk, Rzeszów
  - GASTROMED Sp. z o.o., Torun
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Melita Medical Sp. z o.o., Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - EuroMediCare Szpital Specjalistyczny z Przychodnia, Wroclaw
  - ETG Zamosc, Zamość
- Slovakia (4):
  - FNsP F.D.R. Banska Bystrica, Banská Bystrica
  - Cliniq s.r.o., Bratislava
  - KM Management spol. s r.o., Nitra
  - GASTRO I. s.r.o., Prešov
- Spain (8):
  - Hosp. Gral. Univ. Dr. Balmis, Alicante
  - Hosp Reina Sofia, Córdoba
  - Complejo Hosp Univ. de Ferrol, Ferrol
  - Hosp. Univ. de La Paz, Ferrol
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Madrid
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Hosp. Alvaro Cunqueiro, Vigo
- Taiwan (4):
  - Chang-Hua Christian Hospital, Changhua
  - Far Eastern Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency